CLINICAL TRIAL: NCT05295771
Title: Evaluation of Geistlich Fibro-Gide ® in Comparison to Autogenous Connective Tissue Graft in Gingival Phenotype Modification Prior to Orthodontic Maxillary Expansion.
Brief Title: Evaluation of Geistlich Fibro-Gide ® and Autogenous Connective Tissue Graft Prior to Orthodontic Maxillary Expansion.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit participants.
Sponsor: University of Alberta (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00112336
Record Dates: First submitted 2021-12-23; First posted 2022-03-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Thin Gingiva; Transverse Maxillary Deficiency; Cross Bite
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: 30 patients with bilaterally thin gingival phenotype and minimal keratinized tissues will be treated randomly (left or right maxillary site to be randomized) with either Geistlich Fibro- Gide ® (Test arm) on one side and Autogenous Connective Tissue Graft (Control arm) on the contralateral side of the mouth.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test arm (Experimental): Geistlich Fibro-Gide ®.
  Interventions: Procedure: Gingival Phenotype Modification
- Control (Active Comparator): Autogenous Connective Tissue Graft.
  Interventions: Procedure: Gingival Phenotype Modification

INTERVENTIONS:
Procedure: Gingival Phenotype Modification — Autogenous Connective Tissue Graft is the current gold standard for soft tissue phenotype modification. This is being compared with a substitute material called Geistlich Fibro-Gide ® for soft tissue phenotype modification before orthodontic treatment. Geistlich Fibro-Gide ® is a porcine, porous, resorbable and volume-stable collagen matrix, designed for soft-tissue regeneration. Surgical flap design will be an envelope for both interventions.

SUMMARY:
Teenage children and adults often undergo orthodontic treatment each year to improve their dental esthetics and chewing function. One common problem they present with is having a small maxilla compared to the mandible. The standard of treatment to correct this issue is to expand the maxilla using either a tooth-anchored expander, a bone-anchored expander, or braces. Unfortunately, these treatment options can sometimes result in a loss of gum tissue and supporting structures of the teeth. Certain patients, especially ones that have thin gum tissue, are at a higher risk of this gum tissue loss. Orthodontic treatment for these patients will expand their jaw, causing further pressure on already thin gums. An increasingly common treatment to prevent this is to proactively modify patient's thin tissue surgically prior to their orthodontic treatment so they can withstand the tooth movement. The gold standard of doing this surgical intervention consists of harvesting a connective tissue from the palate which is not well tolerated by the younger population. Our study will evaluate the use of a biomaterial substitute instead of harvesting the patient's own tissue to thicken the gingival tissues. Surgical healing, patient satisfaction, pain index, as well as tissue contour post orthodontic treatment will be assessed thoroughly. This study will help us understand: 1) if biomaterials can be a substitute for traditional autogenous gum grafts to help thicken the patient's gum tissue prior to orthodontic treatment, and 2) if they are able to withstand the pressure of orthodontic movement. This will be the first long-term study of this kind.

DETAILED DESCRIPTION:
This study will be a prospective, single-center, blinded, randomized, split-mouth study. Upon ethics approval from the University of Alberta research information services (ARISE), patients will be recruited from Kaye Edmonton Clinic (KEC). This study evaluates the long-term success of Geistlich Fibro-Gide® in comparison to autogenous connective tissue graft for the treatment of gingival phenotype modification of patients with thin gingiva undergoing orthodontic arch expansion in the KEC Graduate Orthodontics clinic. A total of 30 subjects (n=30) will be enrolled in this study. Sample size was estimated based on 80% power, alpha of 0.025, and results from past studies that have been conducted to detect a 10 to 15% difference in gingival tissue recession post orthodontic treatment with a 15% standard deviation (a patient sample of 25 would be ideal). Given the long-term nature of this study, with normal drop-out rates, 30 subjects will ensure an adequate sample size for effective statistical comparison.

In this study, 30 patients with bilaterally thin gingival phenotype and minimal keratinized tissues as determined by standardized studies will be treated randomly (left or right maxillary site to be randomized) with either Geistlich Fibro- Gide ® (Test arm) on one side, and autogenous connective tissue graft (Control arm) on the contralateral side of the mouth. Regular post-surgical follow-up visits will be conducted at weeks 2, 4, 12, 24, and up to 2 years post orthodontic treatment completion. Since orthodontic maxillary expansion most commonly affects maxillary molars (predominantly mesial root), canines and both premolars, the study will restrict treatment sites to only these teeth. The selection of these teeth will help distinguish directly anchored teeth (molars), having force applied through wire (premolars) and secondary expansion effect (canine). In this interventional study, each patient will be randomly assigned to receive either Fibro-Gide® or autogenous connective tissue graft (split-mouth, parallel assignment). The outcomes examiner will be blinded to the intervention used by the periodontist. The primary outcome will be measured by standardized periodontal charting and gingival measurements recorded in axiUm at each visit during the study. This will include recording clinical attachment levels, periodontal probing, gingival margin level in relation to cemento-enamel junction (CEJ), gingival phenotype class, thickness and width of keratinized tissue, periapical radiographs, and clinical photographs recorded during each phase of the study for comparative analyses. Secondary outcomes will be analyzed by utilizing standardized pain indices and post surgical wound healing assessments as described in previous studies.

Patients eligible to participate in the study will be presented with study details and relevant consent forms. Surgical incision design and suturing will be done in accordance with an envelope technique.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for this study include patients ranging from 13 to 17 years of age requiring maxillary expansion;
* presence of all permanent dentition, presence of unilateral or bilateral cross-bite or transverse maxillary deficiency,
* subjects must have at least one tooth with thin gingival phenotype on maxillary canines, premolars or first molars (mesial root only) on either side;
* teeth should have less than 2 mm of keratinized gingiva to be considered for surgical intervention
* subjects should be systemically health.

Exclusion Criteria:

* Exclusion criteria would include patients with previous orthodontic treatment done,
* patients with Class V restorations or abfractions that obliterate cementoenamel junction
* patients with active caries or endodontically involved teeth
* immunocompromised patients that can influence wound healing
* patients with parafunctional habits
* patient with any history of smoking
* pregnant or lactating females
* teeth that have greater than Miller grade I mobility.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Keratinized Tissue Thickness | Before orthodontic treatment commences on average 4 weeks after surgery.
  The thickness of the keratinized gingiva will be measured on the mid buccal of the tooth 1 mm apical to the gingival margin using an endo- reamer at the site of surgical intervention.
Keratinized Tissue Width | 12 weeks after surgery
  Measure the width from the free gingival margin to the mucogingival junction at the site of surgical intervention.
Keratinized Tissue Width | 24 weeks after surgery
  Measure the width from the free gingival margin to the mucogingival junction at the site of surgical intervention.
Gingival margin level in relation to the Cemento Enamel Junction CEJ | 12 weeks after surgery
  The gingival margin will either be at the CEJ, apical to it or coronal to it at the site of surgical intervention.
Gingival margin level in relation to the Cemento Enamel Junction CEJ | 24 weeks after surgery
  The gingival margin will either be at the CEJ, apical to it or coronal to it at the site of surgical intervention.

SECONDARY OUTCOMES:
Duration of Surgery | Day of surgical intervention
  For both the test and control interventions, the duration of the surgical procedure will be recorded from the time of anesthesia to the time of placing the last suture.
Visual Analog Score for Pain | One day after surgery.
  To assess the level of pain experienced by the patient due to the surgical intervention.
Visual Analog Score for Pain | 2 weeks after surgery.
  To assess the level of pain experienced by the patient due to the surgical intervention.
Visual Analog Score for Discomfort | One day after surgery.
  To assess the level of discomfort experienced by the patient due to the surgical intervention.
Visual Analog Score for Discomfort | 2 weeks after surgery.
  To assess the level of discomfort experienced by the patient due to the surgical intervention.
Wound Healing Index | 2 weeks after surgery.
  To assess the wound healing following surgical intervention using an index given by Huang et al 2005 that scores from 1- 3.
Wound Healing Index | 4 weeks after surgery.
  To assess the wound healing following surgical intervention using an index given by Huang et al 2005 that scores from 1- 3.

CONTACTS AND LOCATIONS:
Overall Officials: Monica P Gibson, BDS,MS(Perio),PhD,FRCD(C), Principal Investigator — U of Alberta Co-Director,Perio Graduate Prog,Faculty of Medicine & Dentistry-Dentistry Dept
Locations (1):
- University of Alberta, Kaye Edmonton Clinic, Edmonton, Alberta, Canada